CLINICAL TRIAL: NCT00122070
Title: Quetiapine Treatment for Symptoms Associated With Borderline Personality Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: David J. Rissmiller, D.O., UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 702787; IRUS QUET 0246
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Personality Disorder; Quetiapine; Atypical Antipsychotics; Seroquel; Antipsychotics
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Quetiapine at dosage of 50 to 150 mg
  Interventions: Drug: Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate — Dosage can vary from 50 to 150 mg at PI's discretion
  Other Names: Seroquel

SUMMARY:
Objective:

The objective of this study is to quantitatively examine the efficacy of Seroquel (active ingredient quetiapine fumarate) in subjects with Borderline Personality Disorder (BPD). A secondary objective is to characterize the safety and tolerability of utilizing quetiapine in patients with Borderline Personality Disorder.

Design:

Investigator initiated, 6-week, non-placebo controlled, non-randomized, open-label, single drug, single-center, medication trial.

Participants:

Volunteers (n = 15) diagnosed with Borderline Personality Disorder using the Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II).

Interventions:

Subjects with Borderline Personality Disorder are washed out of all other medications. The subjects are then given the study drug at a dose within the drug's known therapeutic range.

DETAILED DESCRIPTION:
Study Design: A six week, open-label, flexible dosing study using quetiapine. Subjects who qualify at Screening will then proceed to the baseline visit. If all inclusion and exclusion criteria are met, subjects will be administered quetiapine at the baseline visit. Enrollment will be 15 subjects. Enrollment is expected to last for a 6 month period.

Study Flow Sheet

Duration of Study and Visit Schedule. The subjects will have visits at the following intervals:

* Screening (Day -1 to -14)
* Visit 1 (Baseline)
* Visit 2 (Week 1)
* Visit 3 (Week 2)
* Visit 4 (Week 3)
* Visit 5 (Week 4)
* Visit 6 (Week 5)
* Visit 7 (Week 6)

Screening visit (Day -1 to -14): The following procedures will be performed:

1. Review of Inclusion and Exclusion criteria
2. Informed consent: Subject will be enrolled after signing an IRB approved informed consent. A signed copy will be given to the subject.
3. Review of Concomitant Medications
4. Medical/Disease History & Physical Exam, Vital Signs: The subject will have a H&P administered by an investigator. Weight, TPR, BP will be assessed. This will be done in Family medicine by Dr. Robert Hudrick, DO or Dr. Andrea Woll, DO.
5. A 12 Lead EKG will be done in Family medicine by Dr. Robert Hudrick, DO or Dr. Andrea Woll, DO.
6. Diagnostic Interview and Psychological Testing: Mental status will be conducted by the investigator and a SCID I and SCID II psychological test will be administered for screening and the Beck Anxiety Inventory (BAI), Beck Depression Inventory (BDI-II), Buss-Durkee Hostility Inventory (BDHI), Global Assessment of Functioning (GAF), Symptom Checklist 90 (SCL-90-R) and the Clinical Global Impression Scale (CGI) for severity of illness (Global Improvement and Efficacy not rated) will be utilized to measure the efficacy of quetiapine in this disorder.
7. Lab Parameters: Clinical laboratory samples will be collected and tests will be performed at Kennedy Health System Cherry Hill, NJ. They will be as follows:

   A. Comprehensive Metabolic Panel
   * albumin
   * total bilirubin
   * calcium
   * carbon dioxide
   * chloride
   * creatinine
   * glucose
   * alkaline phosphatase
   * potassium
   * total protein
   * sodium
   * SGOT (AST)
   * SGPT (ALT)
   * urea nitrogen (BUN)

   B. Urine Drug Screen
   * amphetamines
   * barbiturates
   * benzo
   * cocaine
   * opiate
   * PCP
   * cannabinoids

   C. Urine HCG in women

   D. TSH

   E. CBC/Differential

   F. Electrocardiogram: EKG will screen for heart disease and arrhythmias
8. Subjects who have abnormal laboratory results will be discontinued from the study.

Visit 1 (Baseline).

Review of the following:

* Lab work
* Adverse Events
* Concomitant Medications
* Inclusion and Exclusion Criteria
* Beck Anxiety Inventory (BAI)
* Beck Depression Inventory ( BDI-II)
* Buss-Durkee Hostility Inventory (BDHI)
* Global Assessment of Functioning (GAF)
* Symptom Checklist 90 (SCL-90-R)
* Clinical Global Impression Scale (CGI) for severity of illness (Global Improvement and Efficacy not rated)
* Abnormal Involuntary Movement Scale (AIMS)
* Simpson-Angus Scale

Study Medication:

The investigator completes all evaluations and determines the medication dosage.

The study coordinator will then dispense the appropriate number of quetiapine tablets.

Visit 2 (Week 1); Visit 3 (Week 2); Visit 4 (Week 3); Visit 5 (Week 4); Visit 6 (Week 5).

Scales that will be used to assess positive change and medication safety during these visits are:

Scales (in alphabetical order):

* Abnormal Involuntary Movement Scale (AIMS)
* Beck Anxiety Inventory
* Beck Depression Inventory
* Buss-Durkee Hostility Inventory (BDHI)
* Clinical Global Impression (CGI)
* Global Assessment of Functioning GAF
* Simpson-Angus Scale

Inclusion Criteria:

To be considered for inclusion in this study subject must:

* Provide written informed consent before beginning any study related activities
* Be between age 18 and 55 years
* Be able to speak, read and write English and follow simple instructions for completing self-rated scales
* Meet DSM-IV criteria for BPD as assessed by the Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II). Those items screened positive by the subject on the Personality questionnaire will be further evaluated by pertinent subsections of the SKID-II.

Concomitant Therapy

Antipsychotic agents other than quetiapine will not be allowed during the study period. Patients who are taking other antipsychotic medication will require at least a three day washout period prior to the baseline visit.

Patients on anticonvulsants, lithium and benzodiazepines will be allowed to enter the study if they have been on the same dose of these agents for three months prior to the baseline visit

How Will the Study Be Analyzed

Laboratory Studies: Studies will be done at baseline and will screen for liver disease, kidney disease, electrolyte imbalance, thyroid or parathyroid dysfunction, respiratory acidosis or alkalosis, anemia, adequate blood cell and platelet count, pregnancy, and presence of illegal drugs. Any subjects with significant laboratory abnormalities will be excluded from the study.

Adverse Events: Subjects will be screened for the following side effects of quetiapine which are dizziness (10%), postural hypotension (7%), dry mouth (7%), and dyspepsia (6%), tachycardia (7%) and somnolence (18%). Patients will be also be monitored for other rare events including seizures, tardive dyskinesia, and neuroleptic malignant syndrome (NMS). Other less common side effects (> 1%) include headache (19% vs placebo 17%), asthenia (3% vs 2%), abdominal pain (3% vs 1%), back pain (2% vs 1%), fever (2% vs 1%), constipation (9% vs 5%),w eight gain (2% vs 0%), rash (4% vs 3%), rhinitis (3% vs 1%), and ear pain (1% vs 0%).

Data Analysis

The following will be reported and statistically analyzed:

* Number of patients who begin and complete the study (maximum n = 15).
* Patients who dropout of the study or are terminated with reasons.
* Demographic characteristics of the patients.
* Number of patients who had personality disorders in addition to Borderline Personality Disorder.
* The final average dose of quetiapine.
* The total score and percentage change of each scale and subscale utilized in the study and whether there was a statistically significant increase or reduction during the period of quetiapine administration.
* Movement Disorder side effects as assessed by the Abnormal Involuntary Movement Scale and the Simpson-Angus Scale and whether there was a statistically significant increase or reduction during the period of quetiapine administration.
* The number and percentage of adverse events that occurred during the period of quetiapine administration.
* The number and percentage of any abnormal laboratory results that occurred during the period of quetiapine administration.

After completion of data collection, the data will be analyzed to determine appropriate parametric analyses. As the N for this study will be 15, a T-test analysis may be applicable if the data permit. We anticipate a preliminary demonstration of treatment effect. Individual weekly scores will serve as dependent variables which lend themselves to a one-way analysis to demonstrate difference between baseline and 6 weeks of active treatment. If our data permit, a two-way T-test will also be employed to demonstrate statistically significant differences in treatment effect. As our data will likely require the utilization of multiple two-way analyses, our data will be Bonferroni corrected in order to adjust for the possibility of false positive (type II) errors. Other parametric analyses will be employed as the data warrant.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before beginning any study related activities
* Be between age 18 and 55 years
* Be able to speak, read and write English and follow simple instructions for completing self-rated scales
* Meet DSM-IV criteria for BPD as assessed by the Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II).

Exclusion Criteria:

* Are pregnant or lactating.
* Have participated in any other studies involving investigational products within 30 days prior to entry into this study.
* Are undergoing an acute withdrawal syndrome from drugs or alcohol.
* Have an Axis I diagnosis of Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder or Bipolar I Disorder as diagnosed by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I), and pertinent subsequent for ruling out exclusionary diagnoses.
* Have an unstable medical disorder as determined by physical examination or laboratory testing. The primary investigator will be responsible for making this judgment based on the above.
* Had an unsatisfactory response to a previous adequate trial of quetiapine as judged by a study investigator.
* Patients cannot begin psychotherapy during the study period, but may continue if started prior to the study.
* Patients who are currently receiving quetiapine therapy may not undergo a washout period and then restart quetiapine in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist 90 scale (SCL-90-R) | 8 weeks

SECONDARY OUTCOMES:
Safety and tolerability will be measured at Baseline and weekly using the following scales: Simpson-Angus Extrapyramidal Side Effect Scale (SAS), Barnes Akathisia Scale (BAS), and Abnormal Involuntary Movement Scale (AIMS). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Rissmiller, DO, Principal Investigator — University of Medicine and Dentistry of New Jersey - School of Osteopathic Medicine
Locations (1):
- University of Medicine and Dentistry of New Jersey - School of Osteopathic Medicine - Department of Psychiatry, Cherry Hill, New Jersey, United States